CLINICAL TRIAL: NCT04545619
Title: Acute Performance Evaluation of the QDOT Micro™ Catheter Used With nGEN Generator in Treatment of Patients With Atrial Fibrillation.
Brief Title: Performance of QDOT Micro™ Catheter With nGEN Generator for Patients With AFIB.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BWI_2019_09
Record Dates: First submitted 2020-08-18; First posted 2020-09-11 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Paroxysmal and Early Persistent AFIB (Experimental)
  Interventions: Device: QDOT MICRO System

INTERVENTIONS:
Device: QDOT MICRO System — QDOT Micro Catheter with nGEN Generator

SUMMARY:
This workflow study will further evaluate the acute performance and safety of the QDOT MICRO™ catheter in a clinical setting used in combination with nGEN Generator. Subjects will be followed for 7 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with symptomatic paroxysmal or early persistent AF undergoing a catheter ablation procedure through pulmonary vein isolation.
2. Age 18 or older.
3. Signed the Patient Informed Consent Form (ICF).

Exclusion Criteria:

1. If the patient has had a ventriculotomy or atriotomy within the preceding twelve weeks.
2. Presence of a myxoma or an intracardiac thrombus.
3. Presence of prosthetic valves.
4. Presence of active systemic infection
5. Patient with an interatrial baffle or patch
6. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child bearing age and plan on becoming pregnant during the course of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cardiologie de Montréal (Montreal Heart Institute), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- QDOT-nGEN Catheter: Participants with atrial fibrillation (AF) underwent the ablation procedure with the QDOT MICRO catheter used in combination with the nGEN generator with QDOT software module during standard electrophysiology mapping and radiofrequency (RF) ablation procedures.
Period: Overall Study
Arm/Group | QDOT-nGEN Catheter
Started | 40
QDOT nGEN Catheter Inserted | 39
Completed | 39
Not Completed | 1
Not completed — due to equipment challenges | 1

BASELINE CHARACTERISTICS:
Arm/Group | QDOT-nGEN Catheter
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Acute Procedural Success
Description: Number of participants who achieved acute procedural success were reported. Acute procedural success was defined as confirmation of entrance block in all targeted pulmonary veins (PVs) after administration of adenosine/isoproterenol using the nGEN / QDOT Micro Ablation System. The participants without any QMODE+ applications for PVI were considered as a failure.
Time Frame: Up to 104 days
Population: The effectiveness analysis set included all enrolled participants who met all eligibility criteria and had the investigational device inserted and underwent an ablation procedure with the study catheter used in conjunction with QMODE+ and /or QMODE for pulmonary vein isolation (PVI) (RF energy was delivered).
Measure: Count of Participants; unit: Participants
Arm/Group | QDOT-nGEN Catheter
Number analyzed (Participants) | 38
Participants | 37

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with AEs were reported. An AE was any untoward medical occurrence whether or not related to the study device or ablation procedure.
Time Frame: Up to 104 days
Population: The safety analysis set included all enrolled participants who had the investigational device inserted, regardless if RF energy was delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | QDOT-nGEN Catheter
Number analyzed (Participants) | 39
Participants | 9

ADVERSE EVENTS:
Time Frame: Up to 104 days
Description: The safety analysis set included all enrolled participants who had the investigational device inserted, regardless if RF energy was delivered.
Arm/Group | QDOT-nGEN Catheter
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 8/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QDOT-nGEN Catheter (N=39)
Pyrexia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QDOT-nGEN Catheter (N=39)
Headache (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT04545619/Prot_SAP_000.pdf